CLINICAL TRIAL: NCT03193151
Title: Diagnostic and Therapeutic Applications of Microarrays in Liver Transplantation, a Multicenter Study
Brief Title: Diagnostic and Therapeutic Applications of Microarrays in Liver Transplantation
Acronym: INTERLIVER
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Philip Halloran, Distinguished Professor, University of Alberta
Other Study IDs: ATAGC04
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Liver Dysfunction
Keywords: Liver transplant; global gene expression; molecular diagnostics
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy extract containing RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: liver biopsy — 5 mm fragment of liver transplant biopsy taken for clinical indication

SUMMARY:
INTERLIVER is a prospective observational study of the relationship of the molecular phenotype of 300 liver transplant biopsies to the histologic phenotype and the clinical features and outcomes. A segment of a biopsy performed as standard-of-care for indications, or by center protocol, will be used for gene expression study.

DETAILED DESCRIPTION:
The current standard for biopsy-based diagnoses of dysfunction of liver transplants is histology (the Banff system), an arbitrary international empirical consensus based on lesions and rules, similar in principle to the kidney, heart, and lung histology systems. Recent data-driven approaches using molecular and conventional technologies indicate that such systems frequently produce incorrect diagnoses - perhaps 40-50% in abnormal kidney or heart transplant biopsies and even more in lung biopsies, with great potential for harm to patients due to inappropriate treatment.

To address this unmet need and improve diagnostics in the area of organ transplantation, the Alberta Transplant Applied Genomics Centre (ATAGC, University of Alberta) has developed a new diagnostic system - the Molecular Microscope® Diagnostic System (MMDx) that interprets biopsies in terms of their molecular phenotype, and combines the molecular and histopathological features of transplant biopsies, plus clinical and laboratory parameters, to create the first Integrated Diagnostic System. The MMDx, developed first in kidney transplant biopsies because phenotypes are well established, will now be adapted to liver transplant biopsies. The present study will develop a Reference Set of liver biopsies, adapt the MMDx system to assess and report molecular phenotype of liver biopsies; and validate and refine this system in 300 unselected prospectively collected for clinical indications and a standard of care biopsies from North American and European Centers. In addition to demonstrating the real-time feasibility and potential value of this System in patient care, the study will develop and optimize a transparent and user-friendly reporting format to communicate this information to clinicians and obtain detailed feedback to improve its utility.

Thanks to increasing interest and support from participating centers, INTERLIVER has already received 856 biopsies from 740 participants and will extend the Reference Set to 900 biopsies.

ELIGIBILITY:
Inclusion Criteria:

* biopsy for clinical indications

Exclusion Criteria:

* no consent, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to recruit 300 biopsies from liver transplant patients for clinical indications and the standard of care biopsies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assign molecular scores (probability) of T cell mediated rejection, antibody mediated rejection in liver transplant biopsies, in a reference set of 100 biopsies | two years
  Based on the reference set, create molecular classifier that predicts antibody mediated and T cell mediated rejection for next 200 biopsies

SECONDARY OUTCOMES:
Assign in real time (two working days upon biopsy receipt) molecular scores (probability) of T cell mediated rejection and antibody mediated rejection. | 1 year
  The molecular phenotype of a newly acquired sample predicts the histologic and clinical features of this sample when compared to the reference set.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD, PhD, Principal Investigator — University of Alberta
Locations (15):
- United States (8):
  - University of California San Francisco, Transplant Research Unit, San Francisco, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Henry Ford Transplant Institute, Detroit, Michigan
  - Vanderbilt University Medical Center, Vanderbilt Transplant Center, Nashville, Tennessee
  - Baylor University Medical Center, Annette C. and Harold C. Simmons Transplant Institute, Dallas, Texas
  - Transplant Surgery, VCU Medical Center, Richmond, Virginia
  - Division of Transplant Surgery, University of Washington, Seattle, Washington
- Centenary Institute of Cancer Medicine & Cell Biology, Royal Prince Alfred Hospital, Camperdown, Australia
- University of Alberta, Laboratory Medicine and Pathology, Edmonton, Alberta, Canada
- Poland (4):
  - Dep. of Nephrology, Transplantation & Internal Med., Samodzielny Publiczny Szpital Kliniczny im. A. Mieleckiego, Katowice
  - Independent Public Composite Regional Hospital, Szczecin
  - Warsaw Medical University, Jesus the Child Clinical Hospital, Warsaw
  - Warsaw Medical University, Independent Public Clinical Hospital, Warsaw
- Institute for Liver Science, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Result] Madill-Thomsen KS, Gauthier PT, Abouljoud M, Bhati C, Bruno D, Ciszek M, Durlik M, Feng S, Foroncewicz B, Grat M, Jurczyk K, Levitsky J, McCaughan G, Maluf D, Montano-Loza A, Moonka D, Mucha K, Myslak M, Perkowska-Ptasinska A, Piecha G, Reichman T, Tronina O, Wawrzynowicz-Syczewska M, Zeair S, Halloran PF. Defining an NK Cell-enriched Rejection-like Phenotype in Liver Transplant Biopsies From the INTERLIVER Study. Transplantation. 2025 Aug 1;109(8):1367-1382. doi: 10.1097/TP.0000000000005269. Epub 2025 Jan 9. PMID 39780312
- [Result] Madill-Thomsen K, Abouljoud M, Bhati C, Ciszek M, Durlik M, Feng S, Foroncewicz B, Francis I, Grat M, Jurczyk K, Klintmalm G, Krasnodebski M, McCaughan G, Miquel R, Montano-Loza A, Moonka D, Mucha K, Myslak M, Paczek L, Perkowska-Ptasinska A, Piecha G, Reichman T, Sanchez-Fueyo A, Tronina O, Wawrzynowicz-Syczewska M, Wiecek A, Zieniewicz K, Halloran PF. The molecular diagnosis of rejection in liver transplant biopsies: First results of the INTERLIVER study. Am J Transplant. 2020 Aug;20(8):2156-2172. doi: 10.1111/ajt.15828. Epub 2020 Apr 9. PMID 32090446
- [Result] Madill-Thomsen KS, Abouljoud M, Bhati C, Ciszek M, Durlik M, Feng S, Foroncewicz B, Francis I, Grat M, Jurczyk K, Klintmalm G, Krasnodebski M, McCaughan G, Miquel R, Montano-Loza A, Moonka D, Mucha K, Myslak M, Paczek L, Perkowska-Ptasinska A, Piecha G, Reichman T, Sanchez-Fueyo A, Tronina O, Wawrzynowicz-Syczewska M, Wiecek A, Zieniewicz K, Halloran PF. The molecular phenotypes of injury, steatohepatitis, and fibrosis in liver transplant biopsies in the INTERLIVER study. Am J Transplant. 2022 Mar;22(3):909-926. doi: 10.1111/ajt.16890. Epub 2021 Dec 3. PMID 34780106
- [Derived] Halloran PF. Integrating molecular and histologic interpretation of transplant biopsies. Clin Transplant. 2021 Apr;35(4):e14244. doi: 10.1111/ctr.14244. Epub 2021 Feb 17. No abstract available. PMID 33595110